CLINICAL TRIAL: NCT00774943
Title: A Randomized, Double-blind, Placebo-controlled, Ascending, Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 557 in Subjects With Systemic Lupus Erythematosus
Brief Title: A Study of AMG 557 in Adults With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 20060169
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; ICOSL; B7RP-1; Costimulation
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — AMG 557

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- AMG 557 (Active Comparator)
  Interventions: Drug: AMG 557
- Placebo (Placebo Comparator)
  Interventions: Drug: AMG 557

INTERVENTIONS:
Drug: AMG 557 — A total of 4 cohorts will be administered multiple doses of drug or placebo subcutaneously. Dose escalation will take place by cohort.

SUMMARY:
This is a Phase 1, randomized, placebo-controlled, double-blind, dose-escalation study of repeat SC doses of AMG 557 in adults with Systemic Lupus Erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* Before any study-specific procedure, the appropriate written informed consent must be obtained;
* Men and women, between the ages of 18 and 70 years old, inclusive, at the time of randomization;
* Diagnosis of SLE as defined by the most recent ACR criteria, including a positive ANA at screening or documented positive ANA (the titer should be at least 1:80) in the past.
* SLE duration of at least six months, as diagnosed by a physician;
* Stable disease, defined as no change in SLE therapy within the previous 30 days; and, in the opinion of the investigator, no anticipated need for a change in SLE therapy will be required while the subject is enrolled in the study;
* Normal or clinically acceptable ECG (12-lead reporting ventricular rate and PR, QRS, QT, QTc) at screening and Day -1 based on the opinion of the investigator;
* Body mass index from 18 to 40 kg/m2 at screening;
* Able and willing to complete entire study according to study schedule.
* Immunizations up to date, with a minimum of tetanus, diphtheria, pertussis (td/Tdap), pneumococcal (polysaccharide) and influenza (during flu season) vaccinations, as determined by the Principal Investigator.

Exclusion Criteria:

* Positive serology for HIV antibodies, hepatitis B surface antigen or hepatitis C antibodies (confirmed by PCR or RIBA);
* Have had signs or symptoms of a viral, bacterial or fungal infection within 30 days of study randomization;
* Evidence of active or latent tuberculosis as assessed by PPD or Quantiferon testing at screening;
* Have donated blood or experienced a loss of blood >500mL within 4 weeks of randomization;
* History of ethanol or drug abuse within the last one year prior to randomization;
* Evidence of significant renal insufficiency, defined by:

The glomerular fitration rate < 50 mL/min using the Cockroft and Gault equation;

* Evidence of liver disease (eg, serum ALT or AST > 2x upper limit of normal);
* Total WBC <3000 x 106/L;
* Neutrophil count < 1500 x106/L
* Platelet count <75,000 x 106/L
* Hemoglobin <10g/dL
* Any disorder (including psychiatric), condition or clinically significant disease (other than a diagnosis of SLE) that would, by it progressive nature and/or severity, interfere with the study evaluation, completion and/or procedures in the medical judgment of the investigator. This includes any age related co-morbidites such as presence of congestive heart failure, angina, chronic obstructive pulmonary disease, asthma, and malignancies (other than resected squamous and basal cell carcinoma of the skin).
* Presence or history of vasculitis (comprising internal organs or extremities or leading to peripheral neuropathy) within the last 3 years, presence or history of active CNS lupus (defined as seizure disorder, cerebral vascular accident, psychosis ascribed to SLE , encephalitis, meningitis, and myelitis) requiring therapy within the last 3 years;
* Uncontrolled hypertension (Blood pressure > 150/95);
* Poorly controlled diabetes (HbA1c > 8%);
* Any history of granulomatous disease including autoimmune granulomatous vasculitis and sarcoidosis;
* Underlying condition that predisposes the subject to infections (eg, history of splenectomy);
* Any disorder or condition that prevents the subject from providing truly informed consent;
* Prior administration of any other biologic that primarily targets the immune system (eg, Lymphostat-B, TACI-Ig, or CTLA4-Ig) in the past 9 months. This includes prior administration of AMG 557;
* Presence of AMG 557 anti-bodies;
* Prior administration of rituximab > 9 months with CD19+ B cells <5/µL;
* Administration of cyclophosphamide (or any other alkylating agent), cyclosporine, tacrolimus, or sirolimus, or > 100 mg/day prednisone or equivalent in the 6 months prior to randomization;
* Participated in an investigational drug trial involving a monoclonal antibody (not targeting the immune system) within 3 months or 5 half-lives, whichever time period is longer, prior to randomization;
* Participated in any another investigational drug or device trial within the previous 30 days or 5 half-lives, whichever time period is longer, prior to randomization;
* Administration of >10 mg/day prednisone (or equivalent) in the 30 days prior to randomization;
* Known sensitivity to mammalian derived products;
* Unwilling to practice an effective method of double-barrier contraception as determined by the investigator for the duration of the study;
* Positive serum hCG at screening or positive urine hCG on D-1; or females who are currently lactating;
* Known allergies to shellfish or any excipients found in KLH;
* Previous immunization with KLH.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Subject incidence of treatment-emergent adverse events and the incidence of antibodies to AMG 557. | Throughout study period

SECONDARY OUTCOMES:
Serum PK profile of AMG 557 after multiple dose administrations. Biomarkers of pharmacodynamic activity for AMG 557. | Throughout study period

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- United States (11):
  - Research Site, Anniston, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, San Leandro, California
  - Research Site, Danbury, Connecticut
  - Research Site, Miami, Florida
  - Research Site, Michigan City, Indiana
  - Research Site, Manhasset, New York
  - Research Site, Rochester, New York
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Amarillo, Texas
  - Research Site, Dallas, Texas
- Research Site, Newmarket, Ontario, Canada

REFERENCES:
- [Derived] Sullivan BA, Tsuji W, Kivitz A, Peng J, Arnold GE, Boedigheimer MJ, Chiu K, Green CL, Kaliyaperumal A, Wang C, Ferbas J, Chung JB. Inducible T-cell co-stimulator ligand (ICOSL) blockade leads to selective inhibition of anti-KLH IgG responses in subjects with systemic lupus erythematosus. Lupus Sci Med. 2016 Apr 8;3(1):e000146. doi: 10.1136/lupus-2016-000146. eCollection 2016. PMID 27099766
- [Derived] Welcher AA, Boedigheimer M, Kivitz AJ, Amoura Z, Buyon J, Rudinskaya A, Latinis K, Chiu K, Oliner KS, Damore MA, Arnold GE, Sohn W, Chirmule N, Goyal L, Banfield C, Chung JB. Blockade of interferon-gamma normalizes interferon-regulated gene expression and serum CXCL10 levels in patients with systemic lupus erythematosus. Arthritis Rheumatol. 2015 Oct;67(10):2713-22. doi: 10.1002/art.39248. PMID 26138472
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com